CLINICAL TRIAL: NCT03395340
Title: Phase II Study of Topical Ruxolitinib for Cutaneous Chronic Graft Versus Host Disease (cGVHD)
Brief Title: Topical Ruxolitinib for Cutaneous Chronic Graft Versus Host Disease (cGVHD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Forced to close study due to poor recruitment (company withdrew drug support).
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Edward Cowen, M.D., Principal Investigator, National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 180035; 18-AR-0035
Record Dates: First submitted 2018-01-09; First posted 2018-01-10 (Actual); Results first posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-06

CONDITIONS: Graft Versus Host Disease; JNS Kinase; Topical Administration
Keywords: cGVHD; Epidermal; JAK Inhibitor; Skin; JAK-STAT
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib cream (Experimental): Investigational cream to 1 location; vehicle cream to 2nd location
  Interventions: Drug: Ruxolitinib 1.5% cream
- Vehicle cream (Placebo Comparator): Investigational cream to 1 location; vehicle cream to 2nd location
  Interventions: Drug: vehicle cream

INTERVENTIONS:
Drug: Ruxolitinib 1.5% cream — Topical formulation of ruxolitinib, a Janus kinases (JAK) 1/2 inhibitor.
  Other Names: Opzelura
  Arms: Ruxolitinib cream
Drug: vehicle cream — Matching vehicle cream applied as a thin film
  Arms: Vehicle cream

SUMMARY:
Background:

About half the people who have a hematopoietic stem cell transplant using donor cells get Chronic Graft Versus Host Disease (cGVHD). This is chronic graft versus host disease. Immune cells from the donor may see the body tissues in the person as foreign and attack, causing damage. The skin is the most commonly affected organ. Most cGVHD therapies have serious side effects. The cream ruxolitinib inhibits proteins that may play a role in cGVHD.

Objective:

To test the safety and effectiveness of topical ruxolitinib 1.5 percent cream in people with cGVHD of the skin.

Eligibility:

People ages 12 and older with epidermal skin cGVHD

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Skin sample taken (biopsy) to confirm the diagnosis.

At the baseline visit, participants will have:

Skin disease measured with rulers, photographs, and tracing the outline of skin lesions

To complete questionnaires about their symptoms

Blood and urine tests

Some participants will also have a skin biopsy, or total body photographs while they wear only underwear.

Participants will get the ruxolitinib cream and a placebo cream to apply to 2 separate areas of disease. They will do this twice a day for 6 weeks, if they do not have serious side effects. Neither the study team nor the participant will know which area will get ruxolitinib cream and the placebo cream.

Participants will write down:

* When they apply the creams
* Any side effects
* Any medications they take

Most participants will have 4 visits during the 6 weeks they use the creams. Some will have 3 visits and a phone call to see how they are doing. All participants will get a call 4-6 weeks after they stop. Visits include physical exams, blood tests, skin disease measurements, questionnaires, and photos.

DETAILED DESCRIPTION:
Background:

* Chronic graft-versus-host disease (cGVHD) develops in approximately half of individuals who undergo allogeneic hematopoietic cell transplant (HCT) and is the leading cause of non-relapse mortality.
* There are no skin-targeted therapies for cutaneous cGVHD that are directed to the pathogenesis of cGVHD.
* Many inflammatory cytokines involved in the pathogenesis of cGVHD signal through the Janus kinase (JAK)-Signal Transducer and Activator of Transcription (STAT) pathway.
* Systemic JAK inhibitors have been studied in GVHD murine models and in humans with improvement at the cellular and clinical level.
* Topical JAK inhibitors have not been studied in cutaneous cGVHD but have demonstrated the ability to decrease inflammatory markers as well as improve clinical findings of psoriasis.

Objectives:

* To determine the safety and tolerability of topical ruxolitinib 1.5% cream in patients with cutaneous cGVHD with epidermal involvement (non-sclerotic form)
* To determine the efficacy of topical ruxolitinib 1.5% cream in patients with cutaneous cGVHD with epidermal involvement (non-sclerotic form)

Eligibility:

Inclusion:

* Age greater than or equal to 12 years old
* Histologically confirmed epidermal cGVHD (including lichen planus-like, papulosquamous, erythematous) involving at least 2 separate, non-ulcerated sites that can be delineated by body region (e.g., right forearm and left forearm)
* Stable systemic cGVHD treatment including immunosuppressant therapy for 4 weeks prior to enrollment
* Karnofsky or Lansky score greater than or equal to 60%

Exclusion:

* Concurrent use of JAK inhibitors (topical or systemic), fluconazole, or strong Cytochrome P450 3A4 (CYP3A4) inhibitors
* Known hypersensitivity to JAK inhibitors or their components
* Active infection including cytomegalovirus (CMV), Epstein-Barr virus (EBV), human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV)
* Recurrent or progressive malignancy requiring anticancer treatment
* Patients receiving other investigational agents
* Pregnancy

Design:

* This is a Phase II, placebo-controlled, double-blinded study to determine the safety, tolerability and efficacy of topical ruxolitinib in patients with epidermal cGVHD.
* Participants with at least 2 non-ulcerated sites of epidermal cGVHD will apply topical ruxolitinib 1.5% cream to 1 prespecified site and vehicle cream to the second prespecified site twice a day for 6 weeks.
* Safety will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria. Assessments will occur during visits and/or phone follow-up every 2 weeks during treatment.
* Efficacy will be assessed at 6 weeks. The initial surface areas of the 2 target lesions will be measured at baseline, week 2, and week 6 on evaluable patients, with the option for an in-person assessment at week 4. The percent decline in the surface area of the 2 lesions will be determined, and the difference in decline between the 2 lesions will be calculated, expressed consistently as ruxolitinib decline minus placebo decline.
* A skin biopsy and peripheral blood samples will be collected prior to treatment and at week 6 to evaluate the cutaneous immune compartment cellular infiltrate, cytokine profiling, signal transducer and activator of transcription (STAT) phosphorylation, and in situ cGVHD biomarkers.
* Pharmacokinetic studies will be performed at week 2.
* Up to 15 patients will be enrolled to achieve 10 evaluable patients, defined as participants who remain active at the time of the primary endpoint. 10 evaluable patients will provide 80% power to detect whether these paired differences in the changes from baseline are equal to one standard deviation (SD) of the difference of the changes (effect size=1.0) using a two-tailed 0.05 significance level paired t-test. In practice, a Wilcoxon signed rank test may be used instead of a t-test if the differences are not consistent with a normal distribution (p<0.05 by a Shapiro-Wilks test).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically confirmed epidermal Chronic Graft Versus Host Disease (cGVHD) including lichen planus-like, papulosquamous, and erythematous cGVHD with clinical involvement at 2 separate body regions (e.g. right forearm and left forearm).
* Patients must have measurable disease, defined as at least 2 areas of cutaneous, nonulcerated, epidermal cGVHD involvement. Each site must involve at least 0.5% body surface area (1 palm equivalent) and cannot be a site of current or previous nonmelanoma skin cancer (NMSC).
* Stable immunosuppressant or immunomodulatory systemic cGVHD treatment, including phototherapy and extracorporeal photopheresis, for 4 weeks prior to enrollment.
* Age greater than or equal to 12 years. There is no available safety or adverse events data available for children younger than 12 years of age.
* Karnofsky or Lansky greater than or equal to 60
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,000/mcL
  * platelets greater than or equal to 50,000/mcL
  * hemoglobin > 9 g/dL
  * total bilirubin <1.5X institutional upper limit of normal except if known history of Gilbert's disease
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) less than or equal to 5X institutional upper limit of normal
  * creatinine clearance greater than or equal to 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal.
* Willingness to comply with twice daily application of 2 different creams to 2 separate, prespecified sites.
* The effects of ruxolitinib on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients concurrently receiving a Janus kinase (JAK) inhibitor (topical or systemic).
* Patients receiving any other investigational agents.
* Patients concurrently taking oral fluconazole.
* Patients concurrently taking strong Cytochrome P450 3A4 (CYP3A4) inhibitors.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection including Epstein-Barr virus (EBV), Cytomegalovirus (CMV), human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ruxolitinib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib. These potential risks may also apply to other agents used in this study.
* Recurrent or progressive malignancy requiring anticancer treatment.
* Other cancer (except that for which hematopoietic cell transplantation (HCT) was performed) within 2 years of study entry, except nonmelanoma skin cancer or carcinoma in situ of the breast, uterus, or cervix.
* History of cutaneous malignancy at target lesion site.
* Any participant who, in the investigator's opinion, would be unable to comply with study requirements or for whom participation may pose a greater medical risk.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward W Cowen, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi J, Cooper ML, Alahmari B, Ritchey J, Collins L, Holt M, DiPersio JF. Pharmacologic blockade of JAK1/JAK2 reduces GvHD and preserves the graft-versus-leukemia effect. PLoS One. 2014 Oct 7;9(10):e109799. doi: 10.1371/journal.pone.0109799. eCollection 2014. PMID 25289677
- [Background] Spoerl S, Mathew NR, Bscheider M, Schmitt-Graeff A, Chen S, Mueller T, Verbeek M, Fischer J, Otten V, Schmickl M, Maas-Bauer K, Finke J, Peschel C, Duyster J, Poeck H, Zeiser R, von Bubnoff N. Activity of therapeutic JAK 1/2 blockade in graft-versus-host disease. Blood. 2014 Jun 12;123(24):3832-42. doi: 10.1182/blood-2013-12-543736. Epub 2014 Apr 7. PMID 24711661
- [Background] Zeiser R, Burchert A, Lengerke C, Verbeek M, Maas-Bauer K, Metzelder SK, Spoerl S, Ditschkowski M, Ecsedi M, Sockel K, Ayuk F, Ajib S, de Fontbrune FS, Na IK, Penter L, Holtick U, Wolf D, Schuler E, Meyer E, Apostolova P, Bertz H, Marks R, Lubbert M, Wasch R, Scheid C, Stolzel F, Ordemann R, Bug G, Kobbe G, Negrin R, Brune M, Spyridonidis A, Schmitt-Graff A, van der Velden W, Huls G, Mielke S, Grigoleit GU, Kuball J, Flynn R, Ihorst G, Du J, Blazar BR, Arnold R, Kroger N, Passweg J, Halter J, Socie G, Beelen D, Peschel C, Neubauer A, Finke J, Duyster J, von Bubnoff N. Ruxolitinib in corticosteroid-refractory graft-versus-host disease after allogeneic stem cell transplantation: a multicenter survey. Leukemia. 2015 Oct;29(10):2062-8. doi: 10.1038/leu.2015.212. Epub 2015 Jul 31. PMID 26228813
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-AR-0035.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib Cream
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib Cream
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in the Surface Area Measurement of the Target Lesions for Ruxolitinib Treated Versus Placebo Treated Lesions
Description: The surface area will be measured by tracing the lesion on transparency paper and measuring the area from the transparency. Differences in remaining active surface area at 6 weeks from baseline between the treated and placebo sites were compared to calculate efficacy. A decrease in active surface area would signify improvement in skin disease.
Time Frame: Baseline to week 6
Measure: Number; unit: percent change
Groups:
- Ruxolitinib Treated Lesions: Investigational cream to 1 location
  Ruxolitinib 1.5% cream: Topical formulation of ruxolitinib, a Janus kinases (JAK) 1/2 inhibitor.
- Placebo Treated Lesions: Vehicle cream to 2nd location
Arm/Group | Ruxolitinib Treated Lesions | Placebo Treated Lesions
Number analyzed (Participants) | 1 | 1
percent change | -6.35 | -3.81

2. Primary Outcome: Number of Participants With Grade 3 and Grade 4 Adverse Events
Description: Adverse events were measured by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe. Grade 4 is life-threatening.
Time Frame: date on study, up to approximately 2 months and 12 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Cream
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Change in Overall Severity Visual Analog Scale (VAS)
Description: The Overall Severity VAS is a psychometric response questionnaire to measure subjective characteristics or attitudes that cannot be directly measured on a scale of 0-10; a participants assessment of degree of disease activity on the skin. 0=none and 10 = worst imaginable.
Time Frame: Baseline and week 6
Measure: Number; unit: score on a scale
Arm/Group | Ruxolitinib Treated Lesions | Placebo Treated Lesions
Number analyzed (Participants) | 1 | 1
score on a scale
  Baseline | 7.1 | 7.7
  Week 6 | 3.2 | 5.1

4. Secondary Outcome: Change in Pain Visual Analog Scale (VAS)
Description: The Pain VAS is a psychometric response questionnaire to measure subjective characteristics or attitudes that cannot be directly measured on a scale of 0 (no pain) -10 (worst imaginable pain). The participant draws a line on the scale representing how they feel between 0 (none) and 10 (worst). That line is measured and assigned a value. Scores from Baseline and week 6 will be reported. A change is considered a higher number (worsening of disease) or a lower number (improvement of disease) from baseline.
Time Frame: Baseline and week 6
Measure: Number; unit: score on a scale
Arm/Group | Ruxolitinib Treated Lesions | Placebo Treated Lesions
Number analyzed (Participants) | 1 | 1
score on a scale
  Baseline | 0.3 | 0.3
  Week 6 | 0.1 | 0.1

5. Secondary Outcome: Change in Pruritus Visual Analog Scale (VAS)
Description: The pruritus VAS is a psychometric response questionnaire to measure subjective characteristics or attitudes that cannot be directly measured on a scale of 0 (no itching) -10 (worst imaginable itching). Scores from Baseline and week 6 will be reported. A change is considered a higher number (worsening of disease) or a lower number (improvement of disease) from baseline.
Time Frame: Baseline and week 6
Measure: Number; unit: score on a scale
Arm/Group | Ruxolitinib Treated Lesions | Placebo Treated Lesions
Number analyzed (Participants) | 1 | 1
score on a scale
  Baseline | 0.5 | 0.6
  Week 6 | 0.1 | 0.1

6. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve (AUC) of Ruxolitinib
Description: The AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: A pre-dose trough sample will be collected prior to application of the treatment on the day of the follow up visit. After application in clinic, blood samples will be collected at 1 hour, 2 hour and 4 hours.
Population: This outcome measure was not done. Blood was collected for purposes of eventual pharmacokinetic (PK) and pharmacodynamic studies, including AUC but the assay was not developed because the study was not completed and samples were not run. There are no plans to develop the assay, no data was generated for this Outcome Measure.
Arm/Group | Ruxolitinib Cream
Number analyzed (Participants) | 0

7. Secondary Outcome: Total Clearance (CL) of Ruxolitinib
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 6
Population: This outcome measure was not done. Blood was collected for purposes of eventual pharmacokinetic (PK) and pharmacodynamic studies, including total clearance but the assay was not developed because the study was not completed and samples were not run. There are no plans to develop the assay, no data was generated for this Outcome Measure.
Arm/Group | Ruxolitinib Cream
Number analyzed (Participants) | 0

8. Secondary Outcome: Half-Life of Ruxolitinib
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: as for outcome 6
Population: This outcome measure was not done. Blood was collected for purposes of eventual pharmacokinetic (PK) and pharmacodynamic studies, including half-life but the assay was not developed because the study was not completed and samples were not run. There are no plans to develop the assay, no data was generated for this Outcome Measure.
Arm/Group | Ruxolitinib Cream
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Number of Participants With Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence.
Time Frame: Date treatment consent signed to date off study, approximately 2 months and 12 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Cream
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 2 months and 12 days.
Arm/Group | Ruxolitinib Cream
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib Cream (N=1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03395340/Prot_SAP_000.pdf
  • Informed Consent Form: Assent (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03395340/ICF_001.pdf
  • Informed Consent Form: Affected Patient Consent (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT03395340/ICF_002.pdf